CLINICAL TRIAL: NCT06351046
Title: Preventive Interventions for Chronic Pain Worsening
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Novo Nordic Foundation (Other)
Responsible Party: Principal Investigator, Geana P Kurita, Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: NCT05178082_WP3
Record Dates: First submitted 2024-03-27; First posted 2024-04-08 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-04

CONDITIONS: Chronic Non-Cancer Pain
Keywords: Patient Reported Outcome; Virtual Reality; Pain Intensity; Randomized Controlled Trial; Non-pharmacological treatment
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This is an open label randomized controlled trial (RCT), which will be conducted with patients of the Copenhagen Wound Healing Center at Bispebjerg Hospital in Copenhagen (DK). The trial has two arms (1:1) a VRPS group, and a control group (usual care). Participants will be randomly assigned to one of the groups. Assessments will occur at baseline and 2, 6, 9, and 12 months after intervention.
Masking Description: The statistical analysis of the data will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VRPS program (Experimental): VRPS is based on four evidence-based principles of cognitive-behavioral therapy and pain neuroscience education. For this project we have selected relaxation, mindful escapes, pain distraction games, and dynamic breathing modules.The eight consecutive weeks program period of intervention is composed of one initial physical meeting with 1h duration to explain the basis/principles of the virtual tools offered, how the virtual appliance works and should be used, including safety recommendations as calm environment at home, sitting or lying position during use. Groups of maximum 13 patients will be organized. Patients will be instructed to use the equipment at least once a day and it can be used as many times as they wish per day aiming to reduce pain intensity or to avoid pain. Patients will also be asked to keep a diary to register the equipment use during the study period to secure the data.
  Interventions: Device: Virtual Reality-based Pain Self-management program
- Control group (No Intervention): Participants in the control group will not receive any of the interventions. This study will not interfere with medical treatment plan and patients from the three groups can receive other pain treatment prescribed by physician.

INTERVENTIONS:
Device: Virtual Reality-based Pain Self-management program — The VRPS has a variety of modules that can be used for pain management. For this project we have selected relaxation, mindful escapes, pain distraction games, and dynamic breathing modules. All modules were designed to minimize triggers of emotional distress or cybersickness.
  Other Names: VRPS
  Arms: VRPS program

SUMMARY:
This is an open label randomized controlled trial (RCT), which will be conducted with patients of the Copenhagen Wound Healing Center at Bispebjerg Hospital in Copenhagen (DK). The trial has two arms (1:1): A Virtual Reality based Pain Self-management (VRPS) program group, and a control group (usual care). Included will be 44 patients at least 18 years old; fluent in the Danish language; complaint of pain lasting 3 months or more; in average pain intensity score ≥ 3 (numerical rating scale 0 to 10); access to internet; and willing and available to participate in the study. Excluded will be specialized or multidisciplinary pain treatment at baseline; history of epilepsy, seizure disorder, nausea or dizziness, hypersensitivity to flashing light or motion or other diseases that may prevent use of virtual reality equipment; injury to eyes, face or neck.

DETAILED DESCRIPTION:
Considering the need of interventions to improve pain self-management to interrupt the "pain chronification" process and the indications regarding advantages of cognitive behavioral techniques and technologic resources, the purpose of this study is to test a homebased intervention connecting these areas. Here, the effects of a non-pharmacological technique delivered through a virtual reality-based pain self-management program will be tested in patients with non-cancer pain lasting three months or more. The intervention target primarily pain relief by providing pain regulating strategies.

The investigators will test the main hypothesis that participants assigned Virtual Reality-based Pain Self-management program (VRPS) present reduction of pain intensity among other outcomes at 2 months post-intervention as well as after 6-, 9-, and 12-months follow-up when compared to treatment as usual (control group).The primary aim is to investigate the effects of VRPS on worst pain intensity in the last 24h in patients with non-cancer pain lasting 3 months or more at 2 months post-intervention.The secondary aims are to analyze the effects of the intervention on other patient-reported outcomes measures (PROMs), which are pain intensity at follow-ups, pain interference in daily activities, pain catastrophizing, pain acceptance, health-related quality of life, anxiety, depression, perceived change on over-all pain status, use of analgesic medication, and use of health care system among patients with non-cancer pain lasting 3 months or more.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Fluent in the Danish language
* Complaint of pain lasting 3 months or more; in average pain intensity score ≥ 3 (numerical rating scale 0 to 10)
* Access to internet
* Willing and available to participate in the study.

Exclusion Criteria:

* Specialized or multidisciplinary pain treatment at baseline
* History of epilepsy
* Seizure disorder
* History of nausea or dizziness
* Hypersensitivity to flashing light or motion or other diseases that may prevent use of virtual reality equipment.
* Injury to eyes, face or neck that impedes comfortable use of virtual reality equipment.
* Current cancer disease
* Medical diagnosis of depression
* Cognitive dysfunction that interferers with compliance to the study,
* Currently pregnant or planning to become pregnant during the study period
* No access to the internet during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | At baseline, 2 months, 6 months, 9 months and 12 months after intervention
  Pain intensity for worst pain in the last 24h: Brief Pain Inventory to measure pain intensity, from no pain (0) to worst pain ever (10)

SECONDARY OUTCOMES:
Pain intensity and interference in daily activities | At baseline, 2 months, 6 months, 9 months and 12 months after intervention
  Brief Pain Inventory to measure pain intensity from no pain (0) to worst pain ever (10) at follow-ups and interference on general activity, mood, walking ability, work, social relations, sleep, and enjoyment of life
Pain catastrophizing | At baseline, 2 months, 6 months, 9 months and 12 months after intervention
  Pain Catastrophizing Scale, using a 5-point Likert scale ranging from 0 (never) to 4 (always) to assess patterns of negative cognition and emotion in the context of actual or anticipated pain
Pain acceptance | At baseline, 2 months, 6 months, 9 months and 12 months after intervention
  Chronic Pain Acceptance Questionnaire to assess engagement in activity (despite pain), pain willingness, and total pain acceptance score, using a rating scale from 0 to 6. Never true (0) to always true (6)
Health status | At baseline, 2 months, 6 months, 9 months and 12 months after intervention
  patient-generated outcome assessed by the Measure Yourself Medical Outcome Profile (MYMOP2), which measures effects from health care interventions on physical, emotional, or social symptoms/problems. It is problem-specific and includes general wellbeing
Health related quality of life | At baseline, 2 months, 6 months, 9 months and 12 months after intervention
  Physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health using the RAND 36-Item Short Form Health Survey version 1.0. First, precoded numeric values are recoded per the scoring key. All items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.
Anxiety | At baseline, 2 months, 6 months, 9 months and 12 months after intervention
  General Anxiety Disorder - 7 (GAD-7) is commonly used as a measure of general anxiety severity. Measured on a rating scale,- "from not at all" (0) to "almost every day" (3)
Depression | At baseline, 2 months, 6 months, 9 months and 12 months after intervention
  Patient Health Questionnaires scale (PHQ-9) can help track a patient's overall depression severity as well as track the improvement of specific symptoms with treatment. Measured on a rating scale,- from "not at all" (0) to "almost every day" (3)
Use of medication | At baseline, 2 months, 6 months, 9 months and 12 months after intervention
  Medication used (type and quantity) The information collected will refer to the period from patient inclusion to up one year follow-up.
Use of healthcare system | At baseline, 2 months, 6 months, 9 months and 12 months after intervention
  The number of times that he/she used the health care system because of his chronic pain problem and treatment received (pharmacologic, surgical, rehabilitation, etc.). The information collected will refer to the period from patient inclusion to up one year follow-up.
Number of absent days at work | At baseline, 2 months, 6 months, 9 months and 12 months after intervention
  Number of absent days at work because of pain will be asked directly to the patients through the electronic forms. The information collected will refer to the period from patient inclusion to up one year follow-up.

OTHER OUTCOMES:
Satisfaction with the intervention | At baseline, 2 months, 6 months, 9 months and 12 months after intervention
  Satisfaction with the intervention will be asked to the intervention group by general questions about the intervention experienced with answers in a 6-point scale (0=completely dissatisfied to 5= completely satisfied) and there will be space to write comments.

CONTACTS AND LOCATIONS:
Overall Officials: Geana Kurita, PhD, Principal Investigator — Rigshospitalet, Denmark